CLINICAL TRIAL: NCT04978623
Title: Descriptive Analysis of Morphological Aspects of Nerve Fibers in Demyelinationg Polyneuropathies Using HIGH FREQUENCY Ultrasound
Brief Title: Role of High Frequency Ultrasound in Demyelinating Polyneuropathies
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21neuroperiph01
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patient with CIDP: CIDP, is an acquired chronic inflammatory neuropathy characterised by : progressive symmetrical weakness of the proximal and to a lesser extent distal muscles of the lower and/or upper limbs, altered sensitivity and a decrease/abolition of the osteotendinous reflexes. The condition can be relapsing (30% of cases), chronically progressive (60%), or monophasically with total subsequent recovery (10%). Cranial nerve involvement is possible (5-30% of cases). Neuropathic pain as well as respiratory muscle and sub-clinical central nervous system involvement are described.
  Interventions: Other: high frequency ultrasound
- Patient with MMNCB: Patients with MMNCB are at the crossroads between chronic demyelinating neuropathies and motor neuron diseases, the latter for which they constitute a differential diagnosis. The disease usually presents asymmetrically and affects the upper limbs more frequently. The course of the disease is unpredictable, and may be limited to one or two motor nerves or progress to other motor nerves in the contralateral upper limb and possibly the lower limbs. In all cases, the motor deficit is asymmetrical, multi-truncular in distribution, and is usually accompanied by cramps and fasciculations, and eventually by amyotrophy. Osteotendinous reflexes are usually diminished or abolished in the affected areas, but they may also be preserved in the initial attacks. There is no sensory deficit, although some patients occasionally present with paresthesias, and exceptionally with damage to the cranial nerves (especially CN XII).
  Interventions: Other: high frequency ultrasound
- Patient with Anti-MAG: Anti-MAG is a demyelinating neuropathy characterized clinically by a chronic progressive distal and symmetrical predominantly sensory involvement. This neuropathy belongs to the group of symmetrical acquired demyelinating neuropathies (Distal Acquired Demyelinating Neuropathy (DADS)) which is distinguished from PIDC by: 1. an essentially distal and rather sensitive clinical involvement (unlike PIDC which is proximal and distal with predominantily motor involvement); 2. a strong association with a monoclonal gammopathy of the IgM type (67% of DADS vs 22% of PIDC according to Katz et al, 3. a poor therapeutic response to first line of immunosuppressive drugs (in contrast to PIDC which generally responds well). Certain electrophysiological parameters, such as the demonstration of demyelinating damage with accentuated slowing of distal nerve conduction, make it possible to distinguish anti-MAG neuropathy from CIDP.
  Interventions: Other: high frequency ultrasound
- Patient with L-S: Lewis-Sumner syndrome is an acquired demyelinating polyradiculoneuritis characterised by distal asymmetric upper and lower limb weakness and motor dysfunction that develops in adulthood. It is considered a variant of chronic inflammatory demyelinating polyradiculoneuritis. It has a prevalence of 1-9 per 1,000,000. The diagnosis is made with electroneuromyography (ENMG) which shows marked and persistent conduction blocks, in at least two nerves, having an asymmetric topography, mainly affecting the upper limb, outside the usual areas of compression. Lower limb blocks are much rarer (anterior tibial nerve), and are always located below the fibular neck.
  Interventions: Other: high frequency ultrasound

INTERVENTIONS:
Other: high frequency ultrasound — high frequency ultrasound in subgroups of patients with CIDP, anti-MAG, NMMBC and L-S syndrome

SUMMARY:
The use of neuroimaging in the evaluation of neuromuscular pathologies is a promising and rapidly expandinf field. Among the different imaging techniques employed, nerve ultrasound is of particular interest given it's non invasivity, lack of side effects, accesibility and low cost. This exam provides complementary data to electroneuromyography (ENMG), enabeling the physician to visualise the morphological correspondents of electrophysiological abnormalities with a spatial resolution at least as good as MRI.

Chronic Inflammatory Demyelinating Polyradiculoneuritis (CIDP), Multifocal Motor Neuropathy with Conduction Blocks (MMNBC), Lewis and Sumner syndrome (L-S syndrome) and anti-MAG antibody-associated neuropathies (anti-MAG) are among the main chronic inflammatory neuropathies of autoimmune etiology. The diagnosis of these diseases is based on clinical, paraclinical and ENMG examinations. Several recent studies have highlighted the valuable role of ultrasound not only in the diagnosis but also for follow up of patients afflicted by this group of diseases.

However, the current ultrasound imaging techniques does not allow for a detailed study of the internal structure of the nerves. The developement of technologies with improved resolution contribute to further the knowledge in this innovative field and to better understand the pathophysiological mechanisms responsible for initiation and progression of inflammatory nerve disorders.In the Department of Ultrasound at the Nice University Hospital in France the team have at its disposal a high frequency untrasound that the team use to explore the peripheral nervous system.

The scientific hypothesis of this pilot study rests on the premise that demyelinationg neuropathies are a heterogenous group where different types present with different morphological characteristics not only at the level of the nerve as a whole, but also at the level of the nerve fascicles and of the peri- and intra-neural vascular structures. In this respect, high frequency ultrasound allows us to visualise different segments of affected nerves and to obtain morphological details which the team then compare with existing ultrasound data in the literature (high frequency ultrasound: 10-20 MHz). Thanks to this non-invasive and painless technique, the nerve can be rapidly visualised along its entire length in static and dynamic mode. In addition, high frequency ultrasound will give us access to complementary data on the morphology of the soft tissues and the peri- and intra-neural vascular structures which may be useful in shedding light on the underlying pathophysiologycal processes. Another important aspect is the opportunity to make electromyographic and clinical correlations The main parameter The team will study in ultrasound will be hypertrophy, corresponding to an increase in the cross-sectional area of the nerve. the team will also conduct analysis on other less codified parameters, such as epineural and endoneural vascularisation (using the Doppler mode), as well as nerve fascicles anatomy (size, organisation). Identification of different characteristics may be of diagnostic interest in cases where the clinical, paraclinical and ENMG examinations do not allow us to make a diagnostic and therapeutic decision, but it can also prove useful in the follow-up of patients and response to treatment.

This is a descriptive, pilot, mono-centric, multiparametric and retrospective analysis study on patients followed in our centre with a diagnosis of CIDP, NMMBC, L-S syndrom and anti-MAG

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* 18 years of age or older
* Patients with CIDP or NMMBC or definite anti-MAG neuropathy according to the criteria defined by EFNS 2010
* Signing of an informed consent.
* Affiliation or beneficiary of the social security system

Exclusion Criteria:

* Subjects with a medical condition deemed by the investigator to interfere with the proper conduct of the study.
* Positive pregnancy test.
* Pregnant or breastfeeding woman (a urine pregnancy test will be performed for women of childbearing age) A urine The results will be communicated to the patient by a doctor of her choice.
* Persons deprived of their liberty by a judicial or administrative decision;
* Persons hospitalised without consent;
* Persons of full age who are subject to a legal protection measure or who are unable to express their consent.
* Incapacity of the subject to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in this study came to the Nice University Hospital in the Peripheral Nervous System and Muscle (SNPM) department for a consultation in the context of neuropathy. They were diagnosed with CIDP, MMNBC, anti-MAG and L-S and have undergone an ultrasound in addition to standard diagnosis protocol.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Analysis of nerve size using high frequency ultrasound | 24 months
  Size of cross section area (CSA) (mm) mesured in trasversal section of median and ulnar nerves at wrist, elbow and middle arm

SECONDARY OUTCOMES:
correlation between ultrasound data and clinical data | 24 months
  The study of the correlation between ultrasound data (CSA) and clinical data (degree of functional impairment caused by the neuropathy) will be carried out on the basis of motor deficit score obtained by using functional assessment scales and filling in a self-questionnaire: - MRC-score allowing the assessment of the motor deficit. -
correlation between ultrasound data and clinical data | 24 months
  The study of the correlation between ultrasound data (CSA) and clinical data (degree of functional impairment caused by the neuropathy) will be carried out on the basis of sensory deficit score obtained by using functional assessment scales and filling in a self-questionnaire: - INCAT for the evaluation of sensory deficit.
Correlation between ultrasound data and electrophysiological data | 24 months
  The study of the correlation between the ultrasound data and the electrophysiological data will be carried out on the basis of the ultrasound scores obtained at the level of the predefined nerves and observation sites: - Distal latency (in milliseconds);
Correlation between ultrasound data and electrophysiological data | 24 months
  The study of the correlation between the ultrasound data and the electrophysiological data will be carried out on the basis of the ultrasound scores obtained at the level of the predefined nerves and observation sites: - Motor conduction velocity (in m/s);
Correlation between ultrasound data and electrophysiological data | 24 months
  The study of the correlation between the ultrasound data and the electrophysiological data will be carried out on the basis of the ultrasound scores obtained at the level of the predefined nerves and observation sites: - Total and partial conduction block (reduction in the area and amplitude of the global muscle action potential expressed in percentage));
Correlation between ultrasound data and electrophysiological data | 24 months
  The study of the correlation between the ultrasound data and the electrophysiological data will be carried out on the basis of the ultrasound scores obtained at the level of the predefined nerves and observation sites: - Reduction in the amplitude of the global muscle action potential (amplitude in mV)

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No